CLINICAL TRIAL: NCT06840015
Title: Use of Airpod Pros as Assistive Technology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Dr. Linda Thibodeau, Professor, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25-148
Record Dates: First submitted 2024-12-18; First posted 2025-02-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Adult-Onset; Hearing Aids
Keywords: AirPod Pro (AP); Hearing Aids; Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment group (Experimental): AP, HA, ... (Randomized)
  Interventions: Device: Airpod Pro as hearing assistive technology

INTERVENTIONS:
Device: Airpod Pro as hearing assistive technology — All participants will use and evaluate four types of assistive technology: hearing aids, Airpod pro 2nd and 3rd generation, dedicated wireless remote microphones, and Smartphone wireless remote microphone.

SUMMARY:
The goal of this study is to investigate the suitability and effectiveness of the AirPod Pro 2nd and 3rd generation (AP) as hearing assistive technology for individuals with mild-to-moderate hearing loss when listening in noisy environments. Researchers will compare four types of assistive technology: hearing aids (HAs), AP, dedicated wireless remote microphones, and Smartphone wireless remote microphone.

The main questions it aims to answer are:

* Which assistive technology provides the greatest benefit for speech recognition in noisy environments?
* How do these devices impact listening effort, as measured by reaction time in a dual-task activity and changes in pupil size?
* What are participants' preferences for each device based on how easy it is to understand speech and their overall satisfaction? Participants will visit the lab for a single 3-hour session. They will listen to sentences using each device and repeat what they hear. During this task, their reaction times for the secondary task and changes in pupil size will be measured.

DETAILED DESCRIPTION:
A total of 24 participants will be recruited from the Callier Center, local audiology offices, support groups, and senior centers and will first undergo a pure-tone hearing test in a sound booth. The preferred ear tip for the Airpod Pro 3rd generation (AP) will be selected based on participant's comfort, ensuring it passes the ear tip fit test in the iPhone operating system. Similarly, the appropriate ear tip for the receiver-in-the canal Phonak Paradise hearing aid will be selected. The devices will be fit bilaterally and programmed for the individual's hearing loss using the smartphone or computer. Real-ear measurements will be then conducted with both the HAs and the APs to verify that their amplification reaches the The National Acoustic Laboratories non-linear version 2 (NAL-NL2) target level bilaterally (± 5 decibels) for the individual's degree of hearing loss, using Audioscan Verifit 2 (version 4.26.3).

The speech recognition threshold (SRT) at 70.7% will first be measured using the AP and a 2-down-1-up adaptive procedure, adjusting the signal-to-noise ratio (SNR) of babble noise using Hearing in Noise Test (HINT). The sentence will be presented at 65 dBA constant level from Knowles Electronics Manikin for Acoustic Research (KEMAR) with a mouth simulator positioned 1 meter at 0 degrees azimuth. The noise will be presented from the two speakers positioned 1 meter at 90- and 270-degrees azimuth. The participant must repeat the key words correctly. The SNR step size will initially be set to 4 dB for the first three reversals to enable rapid convergence, then reduced to 2 dB to refine the threshold measurement. This procedure will continue until six to eight reversals are obtained to ensure threshold stability. This approach will provide a reliable measurement of the SRT with the AP and allow enough range for improvements to comparison with other assistive technologies.

Next, the participants will complete a dual-task paradigm at the SNR that resulted in 70.7% performance with AP, both without assistive technology and with technology including HA, AP, dedicated wireless remote microphones (DRM), or Smartphone wireless remote microphone (SRM). The target speech will be presented through KEMAR with a mouth simulator positioned 1 meter at 0 degrees azimuth, with babble noise from two speakers positioned 1 meter at 90- and 270-degrees azimuth. The primary task will involve sentence recognition in babble noise using different AzBio sentence lists mentioned above. The secondary task will utilize a working memory task from PALETA (www.paleta.fob.usp.br). While listening to and repeating the AzBio sentence aloud, participants will simultaneously look at the screen, memorize, and click the sequence of colors. Listening effort will be measured by calculating the difference in response time (RT) for the secondary task between the dual-task condition (primary and secondary) and single-task (secondary only) condition.

Following this, the pupil diameter will be measured while participants repeat sentences presented, serving as an additional measure to more reliably assess listening effort under consistent same speaker, SRT and device settings. The AzBio sentence list (Spahr et al., 2012), consisting of 20 sentences, will be used with each assistive technology condition, totaling five sets. Pupil diameter will be captured using the Tobii Pro Lab Analyzer software (version 1.217, Tobii Technology AB, Stockholm, Sweden) positioned 1 meter in front of the participant. This measure will provide two key insights: listening effort and speech recognition ability. We will then compare listening effort and speech recognition with and without each assistive device to determine which assistive technology provides the greatest benefit for speech recognition and listening effort in noisy environments.

Finally, participants will complete a questionnaire to evaluate their experience with each assistive technology. During the pupillometry session, they will rate the difficulty of the sentence recognition task immediately after using each device. At the end of the session, participants will select their preferred assistive technology with the reason for their choice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years.
* Native English speakers.
* Mild-to-moderate hearing loss confirmed by a pure-tone hearing test (average hearing threshold screening 25 to 55 dB HL across octave frequencies from 250 to 8000 Hz).
* Individuals with no prior hearing aid experience for a year.

Exclusion Criteria:

* Normal hearing.
* Hearing loss worse than moderate.
* Neurological, psychiatric, or ophthalmological conditions that might alter the pupil response.
* Non-native English speakers.
* Individuals with prior hearing aid experience more than a year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Speech recognition threshold at 70.7% | The measurement will be conducted immediately following the intervention within the 2-hour single session.
  Speech recognition threshold (SRT) at 70.7% is the noise level at which a person can correctly repeat 70.7% of sentences. Determine the appropriate dB SNR to measure sentence recognition with assistive technologies. It is measured in decibels (dB). Lower values indicate better performance.
Reponse time of secondary working memory task | The measurement will be conducted immediately following the intervention within the 2-hour single session.
  It refers to the amount of time it takes for a participant to react to and complete the secondary working memory task, performed alongside the primary task (speech recognition). This measurement reflects the participant's cognitive processing speed and listening effort. It is measured in seconds (s). Faster values indicate better performance.
Pupil diameter | The measurement will be conducted immediately following the intervention within the 2-hour single session.
  Pupil diameter reflects the motivation to exert effort through physiological mechanisms that maintain homeostasis, making it a reliable indicator of listening effort. It is measured in millimeters (mm). Larger pupil diameters typically indicates greater exerted effort.
Questionnaire | The measurement will be conducted immediately following the intervention within the 2-hour single session.
  Participants are asked to rate how easy it was to understand the speaker with each device. This scale ranges from "Very easy", "Easy", "Ok", "Hard", to "Very hard". They are also asked to select their most preferred device.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Thibodeau, Ph.D., Study Director — The University of Texas at Dallas; Seeon Kim, Ph.D., Principal Investigator — Callier Center for Communication Disorders
Locations (1):
- Callier Center for Communication Disorders, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Don't have plan to share IPD.

REFERENCES:
- [Background] Levitt H. Transformed up-down methods in psychoacoustics. J Acoust Soc Am. 1971 Feb;49(2):Suppl 2:467+. No abstract available. PMID 5541744
- [Background] Nilsson M, Soli SD, Sullivan JA. Development of the Hearing in Noise Test for the measurement of speech reception thresholds in quiet and in noise. J Acoust Soc Am. 1994 Feb;95(2):1085-99. doi: 10.1121/1.408469. PMID 8132902
- [Background] Spahr AJ, Dorman MF, Litvak LM, Van Wie S, Gifford RH, Loizou PC, Loiselle LM, Oakes T, Cook S. Development and validation of the AzBio sentence lists. Ear Hear. 2012 Jan-Feb;33(1):112-7. doi: 10.1097/AUD.0b013e31822c2549. PMID 21829134
- See also: Platform to Assist in the Execution of Dual Task Tests — https://paleta.fob.usp.br/index.php